CLINICAL TRIAL: NCT03211312
Title: Risk Factors and Prediction Model of Elderly Patients With Cardiovascular Diseases Undergoing Teeth Extraction Surgery
Brief Title: Prediction Model of Cardiac Risk for Dental Extraction in Elderly Patients With Cardiovascular Diseases
Status: Completed | Type: Observational
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Shaojun Ma, visiting staff, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Other Study IDs: Shanghai9th
Record Dates: First submitted 2017-07-06; First posted 2017-07-07 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Cardiovascular Diseases; Elderly Patients; Tooth Extraction
Keywords: Cardiovascular diseases; Prediction model; Dental extraction; Elderly patients
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- older people with cardiac diseases: undergoing teeth extraction surgery

SUMMARY:
This study intends to investigate the relevant risk factors of perioperation complications or mortality in older patients with cardiac diseases undergoing teeth extraction surgery and this study aims to quantify the risk factors and then to establish the predictive scoring systems.

Hypothesis:Preoperative parameters could predict postoperative complications.

DETAILED DESCRIPTION:
This study intends to investigate the relevant risk factors of perioperative complications or mortality in older patients with cardiac diseases undergoing teeth extraction surgery and this study aims to quantify the risk factors and then to establish the predictive scoring systems.

We hope that the benefits will include less patients becoming seriously postoperative complications and mortality after teeth extraction surgery.We also hope the information will help doctors understand the preoperative risks better and therefore make better informed decisions.This may also reduce the overall cost of surgery for patients and hospitals.

ELIGIBILITY:
Inclusion Criteria:1.Adults ≥60 years age 2.Males with cardiac diseases 3.Females with cardiac diseases 4.Listed for teeth extraction surgery

-

Exclusion Criteria:

* 1.patient with malignant arrhythmia 2.Age <60 years age 3.Adults with learning disabilities or dementia 4.Patient unwilling/unable to consent 5.Prisoners

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population are all older patients with cardiac diseases undergoing teeth extraction surgery.
Sampling Method: Non-Probability Sample
Enrollment: 833 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
cardiac complications | 7 days
  the cardiac complications during or after dental extraction,such as cardiac events, perioperative SBP ≥180 mmHg, diastolic blood pressure ≥120 mmHg, heart rate ≥120 beats per minute and increase in blood pressure by 20% or above relative to the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: shaojun ma, master, Study Director — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University,School of Medicie
Locations (1):
- Shanghai Ninth People's Hospital,Shanghai Jiao Tong University School of Medicine,Shanghai,China., Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tang M, Hu P, Wang CF, Yu CQ, Sheng J, Ma SJ. Prediction Model of Cardiac Risk for Dental Extraction in Elderly Patients with Cardiovascular Diseases. Gerontology. 2019;65(6):591-598. doi: 10.1159/000497424. Epub 2019 May 2. PMID 31048587